CLINICAL TRIAL: NCT04148573
Title: Randomized, Double-blind, Placebo Controlled, Parallel, Multicentric, Phase IIa Clinical Trial to Evaluate Safety, Tolerability, Therapeutic Efficacy of Daily Oral Treatment NFX88 on Neuropathic Pain in Patients With Spinal Cord Injury
Brief Title: Clinical Trial to Evaluate Safety, Tolerability and Efficacy of NFX88 in SCI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neurofix S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NFX88-2A-2018; 2018-004792-13 (EudraCT Number)
Record Dates: First submitted 2019-06-04; First posted 2019-11-01 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-12

CONDITIONS: Neuropathic Pain; Spinal Cord Injuries
MeSH Terms: conditions — Neuralgia; Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm NFX88 - 1 (Active Comparator): 1.05 g/day NFX88
  Interventions: Drug: NFX88 - 1
- Arm NFX88 - 2 (Active Comparator): 2.10 g/day NFX88
  Interventions: Drug: NFX88 - 2
- Arm NFX88 - 3 (Active Comparator): 4.20 g/day NFX88
  Interventions: Drug: NFX88 - 3
- Arm PLACEBO - 4 (Placebo Comparator): Placebo
  Interventions: Drug: PLACEBO - 4

INTERVENTIONS:
Drug: NFX88 - 1 — 3 times a day
  Other Names: 2OHOA
  Arms: Arm NFX88 - 1
Drug: NFX88 - 2 — 3 times a day
  Other Names: 2OHOA
  Arms: Arm NFX88 - 2
Drug: NFX88 - 3 — 3 times a day
  Other Names: 2OHOA
  Arms: Arm NFX88 - 3
Drug: PLACEBO - 4 — 3 times a day
  Arms: Arm PLACEBO - 4

SUMMARY:
In summary, this small-scale study is designed to demonstrate that the NFX88 is safe and well tolerated, as well as preliminary evidence of improvement in the score of VAS, PD-Q, and PGIC scales.

DETAILED DESCRIPTION:
This is a Phase IIa (proof of concept), randomized, double-blind, placebo controlled, parallel group, multicentric, clinical trial to evaluate the safety, tolerability and efficacy of daily oral treatment with NFX88 in SCI patients who are not receiving opiates or cannabinoids and present neuropathic pain with an average pain score ≥ 4 measured with a VAS scale during the last week at screening

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide written informed consent.
2. Male or Female 18 to 65 years of age.
3. Traumatic complete or incomplete spinal cord injury with C4-T12 level and more than three months since injury. 4. Diagnosed of neuropathic pain with an average pain score ≥

4 measured using the VAS scale during the last week.

5. Stable treatment, for at least 1 month, with pregabalin 150-300 mg/day, that should be maintained at the same dose for 90 days until the end of the study treatment.

6. Normotensive patients defined as patients with blood pressure values between 90-160 for systolic pressure and 50-100 for diastolic pressure.

7. Patients who have been treated with stable doses of neuroactive drugs (antidepressants, anticonvulsants, antispastic and similar medicines) at least during the last month, can also be recruited.

8. Availability for the entire study period, absence of intellectual problems likely to limit the validity of consent to participate in the study or the compliance with protocol requirements; willingness to adhere to the protocol requirements, ability to cooperate adequately, to understand and follow the instructions of the physician or designee.

9. Women who are not postmenopausal (at least 12 months) or surgically sterile must have a negative pregnancy test at screening and at the end of study and either abstain from sexual intercourse or use a highly effective method of birth control for the duration of the study and after 12 weeks after the last dose of study drug.

10. For men: agreement to remain abstinent or use contraceptive measures and agreement to refrain from donating sperm for the duration of the study and after 12 weeks from the last dose of study drug.

Exclusion Criteria:

1. Patients treated with opiates (major and minor) and cannabinoids (synthetic, natural or analogous).
2. Patients with blood pressure higher than those accepted in the inclusion criteria.
3. History of alcohol, drug abuse within 6 months prior to screening.
4. Psychiatric patients or those with moderate or severe cognitive impairment.
5. Patient who is pregnant or lactating.
6. Patient who shows evidence of significant liver or kidney disease, or any other conditions known to interfere with the absorption, distribution, metabolism or excretion of drugs or known to potentiate or predispose to undesired effects.
7. Patient who has clinically significant diseases and/or infections captured in the medical history or evidence of clinically significant findings on physical examination and/or clinically significant ordinary laboratory evaluations (haematology, biochemistry, and urinalysis) or ECG.
8. Patient who is currently participating in another clinical trial of an investigational drug or medical device within 90 days prior to screening.
9. Inability to comply with study protocol.
10. Patient unable to swallow 12 1-gram tablets.
11. History of cancer except local basal or squamous cell carcinoma of the skin that has been excised.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
Incidence of serious adverse events | 90 days
  Safety and tolerability of NFX88 administered for 90 days will be evaluated by assessing the number of AE
Incidence of severity adverse events | 90 days
  Safety and tolerability of NFX88 administered for 90 days will be evaluated by assessing the severity and type of AE
Incidence of specific laboratory abnormalities | 90 days
  Safety and tolerability of NFX88 administered for 90 days will be evaluated by assessing specific abnormalities of laboratory values
Incidence of relevant changes in vital signs | 90 days
  Safety and tolerability of NFX88 administered for 90 days will be evaluated by assessing that there are not relevant changes in vital signs that may affect the safety of the patient
Incidence of relevant changes in 12-lead ECGs | 90 days
  Safety and tolerability of NFX88 administered for 90 days will be evaluated by assessing the ECGs to prove that there are not relevant changes in this test through the trial
No changes in MAS and AIS scales. | 90 days
  Safety and tolerability of NFX88 administered for 90 days will be evaluated by assessing that there are not relevant changes in the MAS (e.g. to monitor spasticity worsening) and ASIA (e.g. to monitor neurological worsening) scores.

SECONDARY OUTCOMES:
Improvement in neuropathic pain scales VAS, PD-Q, and PGIC | 90 days
  Reduction from V1 to EoT in pain intensity in the VAS scale, reduction from SV to EoT in the likelihood of neuropathic pain in PD-Q scale and global improvement at EoT in patient's condition according to the PGIC scale.

CONTACTS AND LOCATIONS:
Overall Officials: ANTONIO OLIVIERO, MD, Principal Investigator — HOSPITAL DE PARAPLEGICOS DE TOLEDO
Locations (7):
- Spain (7):
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Vall de Hebron, Barcelona
  - Instituto Guttmann, Barcelona
  - Hospital Virgen de las Nieves, Granada
  - Hospital los Madroños, Madrid
  - Hospital Virgen del Rocio, Seville
  - Hospital de paraplegicos de Toledo, Toledo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Avila-Martin G, Galan-Arriero I, Ferrer-Donato A, Busquets X, Gomez-Soriano J, Escriba PV, Taylor J. Oral 2-hydroxyoleic acid inhibits reflex hypersensitivity and open-field-induced anxiety after spared nerve injury. Eur J Pain. 2015 Jan;19(1):111-22. doi: 10.1002/ejp.528. Epub 2014 May 13. PMID 24824524
- [Result] Avila-Martin G, Mata-Roig M, Galan-Arriero I, Taylor JS, Busquets X, Escriba PV. Treatment with albumin-hydroxyoleic acid complex restores sensorimotor function in rats with spinal cord injury: Efficacy and gene expression regulation. PLoS One. 2017 Dec 15;12(12):e0189151. doi: 10.1371/journal.pone.0189151. eCollection 2017. PMID 29244816

DOCUMENTS (2):
  • Study Protocol (2018-12-28): https://cdn.clinicaltrials.gov/large-docs/73/NCT04148573/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-08): https://cdn.clinicaltrials.gov/large-docs/73/NCT04148573/SAP_001.pdf